CLINICAL TRIAL: NCT05243732
Title: Music Listening for Psychological and Emotional Wellbeing in Adults With Acquired Visual Impairment: a Feasibility Study
Brief Title: Music Listening for Wellbeing in Adults With Acquired Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1021-07
Record Dates: First submitted 2022-01-07; First posted 2022-02-17 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-05

CONDITIONS: Visual Impairment; Low Vision; Depression; Anxiety; Stress; Emotional Adjustment
MeSH Terms: conditions — Vision Disorders; Vision, Low; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability pre/post-test design
Who Masked: Outcomes Assessor
Masking Description: The participants will be randomised into two groups, mindful music or music listening in a 1:1 ratio using a randomisation software (https://www.randomizer.org/) and block randomisation to ensure equal distribution of groups between age and number of years living with a visual impairment. The researchers who are managing and running the study will not be blinded to the assignment of the groups. The participants will not be blinded to their allocated group, as participants would clearly know if they listened to their own preferred music alone or with mindfulness instructions. However, the researchers will blind the participants from the study hypothesis and which listening group is the control condition to minimise risk of bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Music Listening (Experimental): Participants in the mindful music listening group, will receive personalised music playlists based on music tracks or albums or genres suggested by the participant in the pre-intervention survey. The playlist will be created on the streaming platform they are subscribed to.
  In addition to listening to their preferred music daily, they will be emailed a brief mindful music exercise to complete prior to listening to their preferred music playlist (weeks 1-4). The mindful music exercise will have spoken instructions, and focus on key element of mindfulness of paying attention to the present moment. For example, If participants were to notice any thoughts or sensations arising either during the brief exercise or during subsequent music listening, they are to allow them to pass and to gently bring their attention back to the exercise/music.
  Interventions: Behavioral: Mindful Music Listening
- Music Listening (Active Comparator): Participants in the music listening group will receive personalised playlists based on music tracks or albums or genres suggested by the participant in the pre-intervention survey. The playlist will be created on the streaming platform they are subscribed to. In contrast to the mindful-music condition, no specific listening instructions will be given to the music listening only condition.
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Mindful Music Listening — Participants will be instructed to self-administer this intervention daily, five days a week, for four weeks, 20 to 60 minutes per day at any time that is convenient for them.
  During the intervention period, participants will be recommended to listen to music in a private setting that is quiet, where they will not be disturbed or distracted so they can fully focus on the music.
  Participants in the mindful listening group will be given specific instructions on how to listen and follow mindfulness.
  Arms: Mindful Music Listening
Behavioral: Music Listening — Participants will be instructed to self-administer this intervention daily, five days a week, for four weeks, 20 to 60 minutes per day at any time that is convenient for them.
  During the intervention period, participants will be recommended to listen to music in a private setting that is quiet, where they will not be disturbed or distracted so they can fully focus on the music. No other specific music listening instructions will be given
  Arms: Music Listening

SUMMARY:
A visual impairment (VI) is often associated with reduced psychological wellbeing. Music can be used in a variety of ways to promote psychological wellbeing. Music intervention studies demonstrate that listening to music can provide a distraction from unpleasant thoughts/feelings. Hence, music may serve as a catalyst to improve mood and relieve feelings of depression, anxiety, and stress.

The purpose of this study is to investigate if it is feasible for people with acquired VI to self-deliver daily music listening (music alone or with mindful music listening instructions) for wellbeing, in participants homes, for four-weeks, and to collect data remotely on efficacy in reducing symptoms of anxiety and depression and treatment fidelity.

DETAILED DESCRIPTION:
Detailed Description:

As part of the study participants will be asked to:

* listen to music online at home (for example streaming music using Apple Music, Spotify or the provider participants have an existing account with) for up to one-hour each day, five days a week for four-weeks.
* complete a listening diary log each day (10 minutes duration approximately). This provides an opportunity for participants to record their feelings and emotions after every listening exercise.
* complete surveys to capture evaluative information before and after the four-weeks music listening trial.
* part take in a series of one-to-one consultations via Zoom/MS Teams (video optional) on creating a personalised playlist for each participant, technical and instructional training and follow up progress.
* optional one-to-one interview via Zoom/MS Teams (video optional) on feedback and experience of this daily music listening research study (10 minutes duration approximately).

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Have an acquired vision loss (someone who was not born with vision loss but lost part or all of their vision later in life)
* Have an existing account on a online streaming platform to listen to music
* Own a smartphone/tablet or technology that supports their music streaming platform
* Have the capacity to consent
* Have at least mild symptoms on the Depression Anxiety Stress Scale (DASS-21) screening questionnaire; depression (score: 10 or higher on a scale 0-28+) and/or anxiety (score: 8 or higher on a scale 0-20+) and/or stress (score: 15 or higher on a scale 0-34+)

Exclusion Criteria:

• Anyone who has a hearing impairment that renders the individual unable to listen to music or mindfulness instructions and follow a conversation on the telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | At baseline to Week 5 (Pre to Post intervention)
  Feasibility of the intervention will be reported as the percentage of participants who enrol and complete the entire study.
Attrition rate of the intervention | Week 5 (Post Intervention)
  The percentage of recruited participants dropped out from the study prematurely
To understand the reasons for attrition rate of the intervention | Week 5 (Post Intervention)
  Qualitative methods will be utilised to identify reasons the recruited participants dropped out from the study prematurely via free text comment boxes on the evaluation survey and optional semi-structured interviews.
Acceptability of the intervention | Week 5 (Post Intervention)
  Acceptability will be defined as participant's evaluation of the online intervention using both qualitative and quantitative methods. The acceptability of the intervention will be reported as the percentage of participants who evaluated the intervention and score it 5 being "acceptable" in contrast to 1 being "unacceptable" on a 5-point researcher devised Likert scale. Feedback on the overall intervention will be collated through free text comment boxes on the evaluation survey and optional semi-structured interviews.
Accessibility of the intervention | Week 5 (Post Intervention)
  Accessibility will be defined as participant's evaluation of the online intervention using both qualitative and quantitative methods. The accessibility of the intervention will be reported as the percentage of participants who evaluated the intervention, and score it 5 being "very easy" in contrast to 1 being "very difficult" to use on a 5-point researcher devised Likert scale. To identify the accessibility barriers, free text comment boxes on the evaluation survey will be utilised and optional semi-structured interviews.
Adherence to submission of a music listening diary log | Daily (Week 1 to Week 4)
  Adherence to submission of the music listening diary log will be reported as the percentage of the participants who complete the diary log.
Treatment adherence at 4-weeks from baseline | Week 1 to Week 5 (Pre intervention to Post Intervention)
  Treatment adherence will be reported as the percentage of the participants who complete all aspects of the study, i.e. diary log submissions, all music exercises.
To identify reasons for motivation or barriers to adherence | Week 1 to Week 5 (Pre intervention to Post Intervention)
  Qualitative methods will be utilised to identify reasons for motivation or barriers to adherence using free text comment boxes on the evaluation survey and optional semi-structured interviews.

SECONDARY OUTCOMES:
Changes in Depression levels | Baseline and Week 5 (Pre and Post Intervention)
  Depression will be self-rated by participants using the Hospital Anxiety and Depression Scale (HADS). This is assessed on a scale 0-21, below 7 indicates normal levels, 8-10 means borderline abnormal and 11-21 infers abnormal levels of depression.
Changes in Anxiety levels | Baseline and Week 5 (Pre and Post Intervention)
  Anxiety will be self-rated by participants using the Hospital Anxiety and Depression Scale (HADS). This is assessed on a scale 0-21, below 7 indicates normal levels, 8-10 means borderline abnormal and 11-21 infers abnormal levels of anxiety.
Changes in Stress levels | Baseline and Week 5 (Pre and Post Intervention)
  Stress will be self-rated by participants using the Perceived Stress Scale (PSS-14). This is assessed on a scale 0 to 40. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Nurbanu Somani, MSc MRes BSc, Principal Investigator — Anglia Ruskin University
Locations (1):
- Department of Vision and Hearing Sciences, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafaely L, Carmel S, Bachner YG. Subjective well-being of visually impaired older adults living in the community. Aging Ment Health. 2018 Sep;22(9):1223-1231. doi: 10.1080/13607863.2017.1341469. Epub 2017 Jun 21. PMID 28636409
- [Background] Freeman EE, Munoz B, West SK, Jampel HD, Friedman DS. Glaucoma and quality of life: the Salisbury Eye Evaluation. Ophthalmology. 2008 Feb;115(2):233-8. doi: 10.1016/j.ophtha.2007.04.050. Epub 2007 Jul 26. PMID 17655930
- [Background] Broman AT, Munoz B, Rodriguez J, Sanchez R, Quigley HA, Klein R, Snyder R, West SK. The impact of visual impairment and eye disease on vision-related quality of life in a Mexican-American population: proyecto VER. Invest Ophthalmol Vis Sci. 2002 Nov;43(11):3393-8. PMID 12407148
- [Background] Matthews K, Nazroo J, Whillans J. The consequences of self-reported vision change in later-life: evidence from the English Longitudinal Study of Ageing. Public Health. 2017 Jan;142:7-14. doi: 10.1016/j.puhe.2016.09.034. Epub 2016 Nov 10. PMID 28057201
- [Background] Brown RL, Barrett AE. Visual impairment and quality of life among older adults: an examination of explanations for the relationship. J Gerontol B Psychol Sci Soc Sci. 2011 May;66(3):364-73. doi: 10.1093/geronb/gbr015. Epub 2011 Mar 14. PMID 21402645
- [Background] Rovner BW, Casten RJ. Activity loss and depression in age-related macular degeneration. Am J Geriatr Psychiatry. 2002 May-Jun;10(3):305-10. PMID 11994218
- [Background] Mojon-Azzi SM, Sousa-Poza A, Mojon DS. Impact of low vision on well-being in 10 European countries. Ophthalmologica. 2008;222(3):205-12. doi: 10.1159/000126085. Epub 2008 May 22. PMID 18497531
- [Background] Senra H, Macedo AF, Nunes N, Balaskas K, Aslam T, Costa E. Psychological and Psychosocial Interventions for Depression and Anxiety in Patients With Age-Related Macular Degeneration: A Systematic Review. Am J Geriatr Psychiatry. 2019 Aug;27(8):755-773. doi: 10.1016/j.jagp.2019.03.001. Epub 2019 Mar 7. PMID 31005495
- [Background] Chanda ML, Levitin DJ. The neurochemistry of music. Trends Cogn Sci. 2013 Apr;17(4):179-93. doi: 10.1016/j.tics.2013.02.007. PMID 23541122
- [Background] Bernatzky G, Presch M, Anderson M, Panksepp J. Emotional foundations of music as a non-pharmacological pain management tool in modern medicine. Neurosci Biobehav Rev. 2011 Oct;35(9):1989-99. doi: 10.1016/j.neubiorev.2011.06.005. Epub 2011 Jun 16. PMID 21704068
- [Background] Linnemann A, Ditzen B, Strahler J, Doerr JM, Nater UM. Music listening as a means of stress reduction in daily life. Psychoneuroendocrinology. 2015 Oct;60:82-90. doi: 10.1016/j.psyneuen.2015.06.008. Epub 2015 Jun 21. PMID 26142566
- [Background] Blood AJ, Zatorre RJ. Intensely pleasurable responses to music correlate with activity in brain regions implicated in reward and emotion. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11818-23. doi: 10.1073/pnas.191355898. PMID 11573015
- [Derived] Somani N, Street A, Beukes EW, Zhang J, Allen PM. Music listening for psychological well-being in adults with acquired vision impairment: a feasibility randomised controlled trial. Front Psychiatry. 2025 Feb 25;16:1505283. doi: 10.3389/fpsyt.2025.1505283. eCollection 2025. PMID 40071281

DOCUMENTS (1):
  • Informed Consent Form (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT05243732/ICF_001.pdf